CLINICAL TRIAL: NCT00848211
Title: Phase I/IIA Clinical Study of TUTI-16 in Asymptomatic HIV-1 Infected Subjects
Brief Title: Clinical Study of TUTI-16 in Asymptomatic HIV-1 Infected Subjects
Acronym: THYMON-08001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thymon, LLC (Industry)
Responsible Party: Gideon Goldstein, MD, PhD, THYMON, LLC
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THYMON-08001
Record Dates: First submitted 2009-02-13; First posted 2009-02-20 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections
Keywords: HIV; vaccine; lipopeptide; Tat; TUTI-16; THYMON; Treatment Naive
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- TUTI-16 0.03 mg (Experimental): Subcutaneous injection on Day 0, Day 28, and Day 84
  Interventions: Biological: TUTI-16 (0.03mg)
- TUTI-16 0.1 mg (Experimental): Subcutaneous injection on Day 0, Day 28, and Day 84
  Interventions: Biological: TUTI-16 (0.1mg)
- TUTI-16 0.6 mg (Experimental): Subcutaneous injection on Day 0, Day 28, and Day 84
  Interventions: Biological: TUTI-16 (0.6mg)

INTERVENTIONS:
Other: Placebo — Subcutaneous injection on Day 0, Day 28, and Day 84
  Arms: Placebo
Biological: TUTI-16 (0.03mg) — Subcutaneous injection on Day 0, Day 28, and Day 84
  Arms: TUTI-16 0.03 mg
Biological: TUTI-16 (0.1mg) — Subcutaneous injection on Day 0, Day 28, and Day 84
  Arms: TUTI-16 0.1 mg
Biological: TUTI-16 (0.6mg) — Subcutaneous injection on Day 0, Day 28, and Day 84
  Arms: TUTI-16 0.6 mg

SUMMARY:
This protocol represents the first in human study of TUTI-16, and is being conducted to establish the safety and human immunogenicity (anti-HIV-1 Tat titers) of subcutaneously administered TUTI-16. Activity of TUTI-16 will also be determined in minimizing HIV-1 viral loads and sustaining CD4+ T-cell levels.

DETAILED DESCRIPTION:
HIV-1 Tat protein, a virally encoded toxin, is secreted by HIV-1 infected cells and acts on uninfected cells, rendering them permissive for HIV-1 replication. HIV-1 Tat enhances chronic viral replication and induces immune suppression. Antibodies to Tat inhibit this Tat-mediated transcellular activation in vitro and minimize chronic plasma viremia. HIV-1 Tat activities can be blocked in vitro and in vivo by anti-Tat antibodies.

The Thymon Universal Tat Immunogen (TUTI-16) is a fully synthetic, self-adjuvanting lipopeptide vaccine that is water soluble and administered by subcutaneous injection. In preclinical studies, a priming dose and a three week boost in rats induced a high titer antibody response to the eight known distinct epitope variants of HIV-1 Tat protein. These antibodies block the function of the HIV-1 Tat protein (toxin), which is essential to the maintenance of chronic HIV-1 viremia. Therefore, TUTI-16 has potential as a therapeutic vaccine for HIV-1 in humans.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Age ≥18 and ≤50 years at Screening
* HIV-1 seropositive
* asymptomatic and in generally good health
* no prior anti-retroviral therapy within 6 months of screening
* viral load ≥ 3,000 ≤ 100,000 HIV-1 RNA copies/mL
* CD4+ T-cell count ≥ 400/mm3.

Exclusion Criteria:

* Pregnant/nursing females
* positive for HBV or HCV
* acute Herpetic event
* any clinically significant out-of range laboratory value
* subject is unable or unwilling to discontinue during the study
* participation in another investigational drug/vaccine study within 30 days preceding the first injection of investigational agent in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus A Conant, MD, Principal Investigator — Conant Medical Clinical Research
Locations (1):
- Conant Medical Clinical Research, San Francisco, California, United States

REFERENCES:
- [Derived] Goldstein G, Chicca JJ. Exploratory clinical studies of a synthetic HIV-1 Tat epitope vaccine in asymptomatic treatment-naive and antiretroviral-controlled HIV-1 infected subjects plus healthy uninfected subjects. Hum Vaccin Immunother. 2012 Apr;8(4):479-85. doi: 10.4161/hv.19184. Epub 2012 Feb 16. PMID 22336878

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (0.03mg TUTI-16); Group 2 (0.1mg TUTI-16); Group 3 (0.6mg TUTI-16); Placebo: Subcutaneous injection over the deltoid muscle in the upper arm on Day 0, Day 28, and Day 84
Period: Overall Study
Arm/Group | Group 1 (0.03mg TUTI-16) | Group 2 (0.1mg TUTI-16) | Group 3 (0.6mg TUTI-16) | Placebo
Started | 6 | 7 | 6 | 5
Completed | 6 | 6 | 5 | 5
Not Completed | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (0.03mg TUTI-16) | Group 2 (0.1mg TUTI-16) | Group 3 (0.6mg TUTI-16) | Placebo | Total
Number analyzed (Participants) | 6 | 7 | 6 | 5 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 6 | 5 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44 (10) | 48 (9) | 41 (8) | 51 (5) | 45.9 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 1
  Male | 6 | 7 | 5 | 5 | 23
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 6 | 5 | 24

OUTCOME MEASURES:

1. Primary Outcome: HIV Viral Load
Description: Change in HIV viral load from baseline
Time Frame: baseline and 20 weeks
Measure: Log Mean (Standard Error); unit: HIV RNA copies/mL
Arm/Group | Group 1 (0.03mg TUTI-16) | Group 2 (0.1mg TUTI-16) | Group 3 (0.6mg TUTI-16) | Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 5
HIV RNA copies/mL | -0.18 (0.12) | -0.05 (0.13) | 0.002 (0.11) | 0.26 (0.56)
Statistical Analysis 1: Comparison: Group 1 (0.03mg TUTI-16) vs Group 2 (0.1mg TUTI-16) vs Group 3 (0.6mg TUTI-16) vs Placebo; Test type: Superiority or Other; p = 0.008, ANOVA

2. Secondary Outcome: Determination of Anti-Tat Antibodies
Description: Determination of change in anti-Tat antibody level
Time Frame: baseline and 16 weeks
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Group 1 (0.03mg TUTI-16) | Group 2 (0.1mg TUTI-16) | Group 3 (0.6mg TUTI-16) | Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 5
ng/mL | 20 [20 to 456] | 84 [20 to 181] | 84 [20 to 642] | 20 [20 to 53]

3. Primary Outcome: CD4+ T-cell Count
Description: Change in CD4+ T-cell count from baseline
Time Frame: baseline and 20 weeks
Measure: Log Mean (Standard Error); unit: cells/mm3
Arm/Group | Group 1 (0.03mg TUTI-16) | Group 2 (0.1mg TUTI-16) | Group 3 (0.6mg TUTI-16) | Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 5
cells/mm3 | -65 (48) | -116 (56) | 14 (53) | -59 (22)
Statistical Analysis 1: Comparison: Group 1 (0.03mg TUTI-16) vs Group 2 (0.1mg TUTI-16) vs Group 3 (0.6mg TUTI-16) vs Placebo; Test type: Superiority or Other; p = 0.045, ANOVA

ADVERSE EVENTS:
Arm/Group | Group 1 (0.03mg TUTI-16) | Group 2 (0.1mg TUTI-16) | Group 3 (0.6mg TUTI-16) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 5/6 | 5/7 | 5/6 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (0.03mg TUTI-16) (N=6) | Group 2 (0.1mg TUTI-16) (N=7) | Group 3 (0.6mg TUTI-16) (N=6) | Placebo (N=5)
Headache (Nervous system disorders) | 1 (5) | 0 (0) | 1 (1) | 1 (1)
Injection Site Reaction (General disorders) | 1 (1) | 3 (3) | 3 (8) | 1 (1) — Injection site tenderness, irritation, erythema, pain, induration, swelling
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (4) | 2 (2) — nausea, vomitting, diarrhea, abdominal pain upper
muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (7) | 1 (1) | 0 (0) | 0 (0) — fatigue, myalgia, muscular weakness, arthralgia,

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No